CLINICAL TRIAL: NCT03179059
Title: Resolution of Uncertainty Through Testing: The Impact of Pregnancy Tests on Reproductive and Maternal Health Beliefs and Behaviors in Uganda
Brief Title: Resolution of Uncertainty Through Testing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in field coordination
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of California, San Francisco (Other); Mbarara University of Science and Technology (Other); Ichuli Consulting Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: uganda_study
Record Dates: First submitted 2017-05-24; First posted 2017-06-07 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy Tests
Keywords: Reproductive Health; Family Planning; Randomization Trial; Uganda

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pregnancy tests at baseline & follow-up (Experimental): We offer free pregnancy test service at baseline and at follow-up survey.
  Interventions: Diagnostic Test: Pregnancy test at Baseline; Diagnostic Test: Pregnancy test at follow up survey
- Pregnancy tests only at baseline (Experimental): We offer free pregnancy test service at baseline
  Interventions: Diagnostic Test: Pregnancy test at Baseline
- Do Not Offer Pregnancy Test (No Intervention): Control group. No intervention is implemented.

INTERVENTIONS:
Diagnostic Test: Pregnancy test at Baseline — Among respondents who are randomly selected to receive a free home pregnancy test service, they will be offered the chance to take the test in the presence of the enumerator. Specifically, this would mean they would be given a cup to collect a sample of urine. The respondent would do so privately, then bring the cup back to the enumerator who would dip the home pregnancy tests and assist with interpreting the result. However, respondents can decline to take the test with the enumerator. Treatment assignment will be stratified by whether respondent use modern family planning at baseline.
  Arms: Pregnancy tests at baseline & follow-up; Pregnancy tests only at baseline
Diagnostic Test: Pregnancy test at follow up survey — We will provide a free pregnancy tests in for the future use, they are randomly selected from intervention #1 treatment group.
  Arms: Pregnancy tests at baseline & follow-up

SUMMARY:
Given the high rate of delayed adoption of antenatal care (ANC), and high rates of unintended pregnancy and unsafe abortion in Uganda, research on the period of time before confirmation of pregnancy is critical to understand underlying beliefs that guide behaviors ultimately important for maternal and neonatal health (UDHS, 2011; Hussain, 2013).

Home pregnancy tests - which now cost less than 10 cents each - have the potential to facilitate FP uptake and significantly improve reproductive, maternal and child health outcomes in sub-Saharan Africa, including Uganda. These tests are easy to administer, disposable, inexpensive, and have a low false positive rate. Yet, for women living in rural areas in sub-Saharan countries, these tests are typically unavailable outside of health centers or they are prohibitively expensive.

This study will investigate women's underlying beliefs about pregnancy status and examine how providing access to home-based pregnancy tests - thus facilitating earlier resolution of uncertainty of pregnancy status - influences such beliefs and decisions to take up family planning (FP) or seek appropriate pregnancy services.

The results will inform the design of a larger study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35
* Live in the catchment area

Exclusion Criteria:

- Currently attending school

End Survey if

* Women in menopause
* Women with sterilization
* Women with husband/partner with sterilization
* Women who do not understand what menstrual period is

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
Binary measures for the family planning take up | At end line survey, half a year after intervention
  Use of any modern family planning method, use of oral contraceptives, use of injectables, use of short-acting reversible methods, use of long-acting reversible methods. We will measure take up as binary variables. We will also conduct sub-group analyses among women who are not using modern family planning at baseline and among women who are using modern family planning at baseline

SECONDARY OUTCOMES:
Binary measure of purchase of pregnancy test kit by price | At end line survey, half a year after intervention
  Binary measures for the purchase of pregnancy test kit after baseline. Demand for pregnancy test kit is computed by Becker-DeGroot-Marschak (BDM) or/and Take it or leave it (TIOLI) method. We will also conduct sub-group analyses among women who are not using modern family planning at baseline and among women who are using modern family planning at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ichuli Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No